CLINICAL TRIAL: NCT05335473
Title: Phase I b/ II Clinical Study of Iribrine Mesylate Plus Tucidinostat in the Treatment of HR+/HER2- Locally Relapsed or Metastatic Breast Cancer After Previous CDK4/6 Inhibitor Failure
Brief Title: Iribrine Plus Tucidinostat in the Treatment of HR+/HER2 Advanced Breast Cancer After CDK4/6 Inhibitor Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief Physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-MBC07; CSIIT-C28 (Other: CS)
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: HR Positive HER2 Negative Advanced Breast Cancer
MeSH Terms: interventions — eribulin; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eribulin plus Tucidinostat (Experimental): phase 1b： 3+3 trial design will be used for Tucidinostat dose escalation cohorts phase 2: Eribulin+Tucidinostat
  Interventions: Drug: Eribulin and Tucidinostat

INTERVENTIONS:
Drug: Eribulin and Tucidinostat — phase 1b： 3+3 trial design will be used for Tucidinostat dose escalation cohorts phase 2: Eribulin+Tucidinostat

SUMMARY:
To explore the safety and efficacy of Eribulin plus Tucidinostat amine in patients with HR+/ HER2-advanced metastatic breast cancer

DETAILED DESCRIPTION:
To explore the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) and Phase II recommended dose (RP2D) of the regimen of Eribulin plus Tucidinostat , and to initially explore the safety and efficacy of Eribulin plus Tucidinostat amine in patients with HR+/ HER2-advanced metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

-

Subjects must meet all of the following criteria to be enrolled:

1. Age ≥18 years and ≤75 years at the time of signing the informed consent; 2. The physical status score of the Eastern Oncology Consortium (ECOG) was ≤2 points; 3. Confirmed by pathology as HR+/HER2- (according to American College of Clinical Oncology/American College of Pathologists guidelines) (Note: HER2 feminine is defined as ①IH0; IHC1+; Locally advanced or metastatic IHC2+ : FISH-) Sexual female breast cancer patients, not suitable for radical treatment of the purpose of surgery or radiotherapy; 4. Proving that endocrine therapy is difficult to treat or resistant to endocrine therapy; 5. Used 1-2 chemotherapy regiments in the advanced stage; 6. Received at least one taxane and CDK4/6 inhibitor (including unmarketed ones) at any stage; 7. If a patient in the early stage relapses within 12 months of adjuvant chemotherapy (new), it can be counted as one advanced chemotherapy line Number; 8. The total number of treatment lines in the late stage ≤3 lines; 9. At least 1 measurable lesion was present according to RECIST1.1; External radiation therapy (EBRT) or local area treatment (such as radiofrequency ablation) of the lesion must show evidence of disease progression (according to RECIST 1.1), can be used as target lesion; 10. Life expectancy ≥3 months; 11. The functional level of the organ must meet the following requirements:

1. Blood routine: ANC≥1.5×109/L (no growth factor used within 14 days); PLT 100 x 109 or higher/L (within 7 daysNo corrective treatment was used); Hb≥100 g/L(no corrective treatment was used within 7 days);
2. Blood biochemistry: TBIL≤1.5×ULN; ALT and AST≤3 x ULN; Glutamine transpeptidase GGT≤2.5×ULN; If liver metastasis exists, ALT and/or AST≤5×ULN; Glutamine transpeptidase GGT≤5×ULN; Urea, urea nitrogen (BUN), creatinine (Cr) ≤1.5×ULN;
3. Cardiac color ultrasound: LVEF≥50%;
4. 12-lead electrocardiogram: QT interval (QTcF) corrected by Fridericia method for male <450ms, female<470 ms.

11. The time interval between the end of the last antitumor therapy and the first administration of the study drug meets the following requirements: surgery The interval must be ≥4 weeks (minor surgery, such as tumor biopsy, thoracopuncture, or intravenous catheter placement, is not limited); Recovery of adverse reactions to previous antitumor therapy (radiotherapy, chemotherapy, targeting) to ≤ Grade 1 (phase Ib required patients A washout period of 7-14 days after natural recovery without symptomatic drugs or symptomatic treatment).

12. Voluntarily agrees to and signs a written informed consent and is willing and able to comply with all aspects of the test protocol,The patient may withdraw consent at any time without prejudice to his rights and interests.

Exclusion Criteria:

-

Subjects will not be enrolled if they meet any of the following criteria:

1. Receiving neoadjuvant or adjuvant therapy containing Iribulin within one year prior to treatment initiation;
2. Patients with recurrent or metastatic breast cancer who have failed or responded to previous treatment with Iribulin (achieved CR/PR/SD), but tumor progression within 6 months after cessation of aribulin therapy;
3. Patients who have received any HDAC inhibitor at any time in the past;
4. Participated in clinical trials of unmarketed drugs within 4 weeks before enrollment;
5. Exclude subjects with brain or subdural metastases. Unless the patient has completed local treatment and is stable on imaging Those who had maintained the condition for at least 4 weeks, had stopped systemic sex hormone therapy and had stable symptoms for at least 4 weeks were included(By comparing head enhancement CT or MRI performed during screening with head enhancement performed at least 4 weeks earlier CT or MRI to determine the stability of the lesion);
6. Before screening, the toxicity of the original treatment regimen had not recovered, and there were still more than grade 1 toxic reactions (CTCAE5.0);
7. Clinically significant gastrointestinal abnormalities that may affect drug intake, transport, or absorption (e.g., inability to swallow,Chronic diarrhea, intestinal obstruction, etc);
8. Severe/uncontrolled disease or active infection;
9. Severe cardiovascular injury (greater than NYHA Class II congestive heart failure) History), unstable angina pectoris or myocardial infarction within the past 6 months, or severe arrhythmia;
10. Subjects with allograft requiring immunosuppressive therapy.
11. Subject has active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA≥500 IU/ml; cLiver reference: HCV antibody positive and HCV virus copy number > upper limit of normal); Known human immunodeficiency disease Hiv-positive subjects.
12. Had other malignancies within the previous 5 years, excluding cured papillary thyroid carcinoma and in situ cervix Carcinoma, skin basal cell carcinoma or skin squamous cell carcinoma;
13. Subjects with hypersensitivity to softin B and/or softin B chemical derivatives.
14. Pregnant and lactating women, fertile women who have tested positive for baseline pregnancy tests,or were unwilling to use effective contraception throughout the trial period and within 90 days after the last administration of the study drug age patients;
15. The investigator considers the subject unfit for any medical condition to enter the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
DLT for phaseⅠb | 1 year
  Dose-limiting toxicity defined as any Grade 4 hematological toxicity and any > Grade 3 non-hematologic toxicity.
Progression-Free Survival (PFS) for phase Ⅱ | 2 years
  PFS is defined as the time from the date of treatment to the first date of disease progression or death from any cause.
MTD for phaseⅠb | 1 year
  Maximum tolerated dose is highest dose level in which 6 patients treated with at most 1 experiencing DLT.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) for phaseⅠb | 2 years
  PFS is defined as the time from the date of treatment to the first date of disease progression or death from any cause.
adverse events (AE) | 2 years
  The level of the adverse event (AE) is analyzed according to the Common Terminology Criteria for Adverse Event (CTCAE) (version 5.0).
Objective Response Rate (ORR) | 2 years
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1). The percentage of patients who achieved CR and PR was defined as objective response rate (ORR)
Clinical Benefit Rate (CBR) | 2 years
  CBR is defined as the rate of patients who achieved complete response, partial response, and stable disease for >= 24 weeks as the best response of treatment.
Duration of Response (DOR) | 2 years
  DOR is defined as the time from the date of the first response (≥PR) that is subsequently confirmed to the date of first confirmed disease progression or death, whichever happens first
Overall Survival (OS) | 2 years
  OS defined as the time from the first study treatment administration to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No